CLINICAL TRIAL: NCT05036200
Title: Efficacy, Tolerance and Acceptability of Pulsed Dye Laser on Telangiectasias of the Face and Neckline in Systemic Scleroderma: a Prospective Single-center Open-label Study of 21 Patients
Brief Title: Pilot Study to Evaluate the Interest of PDL in the Management of Telangiectasia of the Face and Neckline in Systemic Scleroderma
Acronym: PDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-065
Record Dates: First submitted 2021-07-19; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Telangiectasia
MeSH Terms: conditions — Telangiectasis | interventions — Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- four pulsed dye laser sessions were administered every eight weeks in the 21 patients (Experimental)
  Interventions: Device: pulsed dye laser

INTERVENTIONS:
Device: pulsed dye laser — four pulsed dye laser sessions were administered every eight weeks in the 21 patients

SUMMARY:
This single-center, prospective, open-label, quasi-experimental, intra-individual comparative study will include a consecutive cohort of 21 patients with diffuse or limited, minimally active scleroderma with 3 to 30 years of evolution.

Patients will have 4 sessions of pulsed dye laser 595 nm spaced 8 weeks apart. The final quadruple evaluation by several evaluators will be 2 months after the last session, on the following criteria: evolution of the number of telangiectasia; subjective improvement score (LINKERT scale); impact on quality of life (SKINDEX score); visual analog pain scale (VAS); adverse events (AEs), including discontinuation of treatment due to post-session purpura (AT-PPS); patient satisfaction (yes or no).

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of pulsed dye laser treatment on facial and neckline telangiectasias in systemic scleroderma by comparing the mean number of telangiectasias.

Secondary Objectives:

Evaluation of the aesthetic efficacy by the patient, observer and adjudication committee Evaluation of the impact on the quality of life after treatment (skindex) Evaluation of treatment tolerance in terms of pain (VAS) and adverse events (purpura, oozing, hyperpigmentation, hospitalization)

ELIGIBILITY:
Inclusion Criteria:

* patient followed in dermatology and/or internal medicine at the University Hospital of Caen for systemic scleroderma
* patient with telangiectasias related to scleroderma
* patient with an aesthetic prejudice

Exclusion Criteria:

* Patient with previous laser treatment for facial telangiectasias.
* Tanned, irritated or traumatized facial skin
* Patient not affiliated to the Social Security system
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the decrease in the number of telangiectasia | baseline and two months after last intervention

SECONDARY OUTCOMES:
Assessment of quality of life after pulsed dye laser treatment using the SKINDEX questionnaire | baseline and two months after last intervention

OTHER OUTCOMES:
evaluation of the aesthetic improvement with an improvement score scored using a LIKERT scale from -1 to +2: from -1= worse; 0= unchanged ; +1= improved ; +2= much improved | baseline and two months after last intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mayo TT, Khan F, Hunt C, Fleming K, Markus R. Comparative study on bruise reduction treatments after bruise induction using the pulsed dye laser. Dermatol Surg. 2013 Oct;39(10):1459-64. doi: 10.1111/dsu.12293. Epub 2013 Jul 30. PMID 23899131
- [Background] Yalcinkaya Y, Pehlivan O, Omma A, Alpay N, Erer B, Kamali S, Ocal L, Inanc M. The relationship between nailfold capillaroscopic assessment and telangiectasia score with severity of peripheral vascular involvement in systemic sclerosis. Clin Exp Rheumatol. 2015 Jul-Aug;33(4 Suppl 91):S92-7. Epub 2015 Mar 23. PMID 25797836